CLINICAL TRIAL: NCT01621698
Title: Early Versus Late Paravertebral Block for Analgesia in Video Assisted Thoracoscopic Lung Resection.
Brief Title: Study of Use of Paravertebral Blocks for Pain Relief in Video Assisted Lung Surgery
Acronym: ErLaPara
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Bristol and Weston NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AN/2012/4036
Record Dates: First submitted 2012-06-08; First posted 2012-06-18 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-09

CONDITIONS: Lung Tumour; Lung Metastases
Keywords: VATS; Paravertebral blocks.; Thoracoscopic surgery.; Analgesia.
MeSH Terms: conditions — Lung Neoplasms; Agnosia | interventions — Saline Solution; Propofol; Fentanyl; Atracurium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early paravertebral block (Active Comparator): The early group will have Local anaesthetic placed at the start of surgery and have normal saline placed at the close.
  Interventions: Procedure: Early paravertebral block
- Late paravertebral block (Active Comparator): The late group will have normal saline placed at the start of surgery and local anaesthetic placed at the close.
  Interventions: Procedure: Late Paravertebral block.

INTERVENTIONS:
Procedure: Early paravertebral block — In this group the local anaesthetic will be injected at the start of surgery soon after incision and normal saline at the end. These will be double blinded.
  Other Names: Bupivicaine; Normal Saline; Propofol.; Fentanyl.; Atracurium.
  Arms: Early paravertebral block
Procedure: Late Paravertebral block. — In the late group local anaesthetic will be injected at close of surgery with normal saline at the start. This will be double blinded.
  Other Names: Bupivicaine; Normal Saline; Propofol.; Fentanyl.; Atracurium.
  Arms: Late paravertebral block

SUMMARY:
This project involves looking at the timing of providing pain relief for patients who are having lung surgery via the use of a small camera inserted into the chest with a scope (Video assisted thorascopy). This procedure can be the source of intense pain both immediately after the procedure and in the longer term leading to chronic pain problems.

Local anaesthetic placed in the paravertebral space which is located adjacent to the spinal column, where the pain nerve fibres are located, is a well recognized method of providing pain relief for these procedures. It is currently unclear as to the best timings for providing this type of pain relief with some centres placing the local anaesthetic at the start of the procedure and some at the end. Placing a high volume of local anaesthetic into this area at the start of the case may provide better short and long term pain relief than placing it at the end of the procedure. The investigators hope to show a difference between the two timings to allow for better pain relief for these procedures. This would be a feasibility study that would lead onto a multicentre trial to eventually create a best practice protocol for pain relief for lung resection via this surgical method.

DETAILED DESCRIPTION:
All patients will receive a general anaesthetic for their VATS procedure with full AAGBI monitoring and the WHO surgical safety checklist will be performed appropriately prior to skin incision. Induction of anaesthesia will be standardised by using propofol and the patient will be paralysed using the muscle relaxant atracurium. The amount given will be at the anaesthetist's discretion and dependent on the patient. Fentanyl at 2.5 mcg/kg will be used at induction of anaesthesia.

A double lumen endotracheal tube will be placed so lung isolation can be performed when necessary for the surgery. Anaesthesia will be maintained using a volatile agent or a target controlled infusion of propofol depending on the preference of the anaesthetist. The patient will be positioned laterally with the operative side up. All patients will receive simple intra-operative analgesia in the form of 1 gram of intravenous paracetamol and diclofenac unless the patient is over 70 or has abnormal renal function. Extra opioid analgesia will be given as intravenous morphine and this will be titrated by the anaesthetist. The amount given will be documented as part of the trial data.

Patients will be warmed to maintain a temperature between 36 and 37 degree Celsius using a warming blanket and warmed intravenous fluids. Anti-emetics in the form of ondansetron 4 mg and dexamethasone 4 mg will also be given unless there are any contraindications.

Prior to surgical incision patients in both groups will receive 1mg/kg 0.25% bupivicaine divided into 3 PV injections between the fifth and tenth thoracic vertebrae. Only trained anaesthetists with experience of over 30 PV insertions will perform the injections. The landmark technique for these injections is as follows: The spinous process of the thoracic vertebra is palpated by the anaesthetist, a 20 gauge needle is inserted 2.5 cm lateral to this and is advanced perpendicularly to the vertical and sagittal planes until the transverse process is contacted. The needle is then walked off the superior border of the transverse process, advanced a further 1 cm and one third of the weight determined local anaesthetic is delivered after careful aspiration.

Both groups will have a PV catheter placed at the start of the procedure and a bolus given straight away. As this is a double-blinded trial the anaesthetist will not know whether the bolus is local anaesthetic or saline solution.

Pharmacy at the research site will provide the 2 premade syringes that will contain either local anaesthetic or saline. The contents of the syringe will be unknown to the anaesthetist as the label will be simply numbered as 1 and 2 to be given in order as the early (1) or late (2) bolus. If it is clinically required to obtain information on what has been given a record will be immediately available from pharmacy. The syringes will be made up as neat 0.25% bupivicaine or 0.9% Normal Saline solution. The equivalent volume of 1mg/kg 0.25% bupivicaine will be injected as a bolus.

Both groups will also receive a 0.25mg/kg 0.25% bupivicaine intercostal block at closing and an infusion of 0.1% bupivicaine will then be commenced at 20mls/hr to continue over the post operative period. Intra-operatively the amount of local anaesthetic given will be under the maximum dose of 2 mg/kg. The maximum dose will not be reached even when the infusion commences due to the fact that time will have passed.

The primary outcome measures that will be used are to review pain scores using VAS on coughing. This will start at arrival in recovery room, which will be described as time zero. It will then be reviewed at time 1,2,4,6,12 and 24 hours. The pain scores are routinely measured by the nurses after this type of surgery, the only difference for the study will be that these scores are measured more often, a timer will be placed with the patient to indicate when the scores should be taken.

Secondary outcome measures will include morphine consumption, which will be noted peri-operatively then again at the time intervals described above. These will be recorded by the recovery staff initially and then continued by the ward nurses with the support of the research team.

Other secondary outcomes measured will include cortisol levels the following day, which will allow review of the neuroendocrine response. The patient will have routine blood tests the morning after the surgery; the cortisol level will be added to this test so the subject will not have extra blood taken. Patient satisfaction scores will be recorded in the form of a questionnaire and will be recorded on the first 2 post-operative days. The length of hospital stay, readmission at 30 days, survival at 30 days and infection rates will also be noted.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be recruited from patients admitted for elective VATS for lung resection.
* Patients aged 18 and over.
* Patient's will be ASA 1,2 or 3.

Exclusion Criteria:

* Patient refusal.
* Emergency surgery.
* Patient unable to provide consent.
* Infection in paravertebral space.
* Patients who attend a chronic pain clinic on high doses of opiate drugs.
* History of Anaphylaxis/allergy to local anaesthetic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Pain score on coughing using Visual Analogue Scale (VAS). | 24 hours.
  Pain scores in first 24 hours to be analysed using area under the curve.

SECONDARY OUTCOMES:
Morphine consumption | 24 hours
  Amount of morphine used in first 24 hours via patient controlled analgesia.
Cortisol levels | 24 hours
  Cortisol measured at routine blood tests after 24 hours.
Length of hospital stay | 3 days (Average)
  Patient's will be followed up for the duration of hospital stay, an expected average of 3 days.
Patient satisfaction scores | 24-48 hours
  Performed using questionnaires.
Readmission rates | 30 days
Survival | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Kajan Kamalanathan, BMBS, Principal Investigator — United Hospitals Bristol NHS Foundation Trust
Locations (1):
- United Hospitals Bristol NHS Foundation Trust, Bristol, United Kingdom